CLINICAL TRIAL: NCT01092351
Title: Open Label Study on the Bacteriological and Clinical Efficacy and Safety of a Nitrofurantoin Formulation Given Twice Daily (Bid) for Seven Days in Uncomplicated Urinary Tract Infection in Adults
Brief Title: Efficacy and Safety of Nitrofurantoin in the Treatment of Uncomplicated Urinary Tract Infections in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mepha Ltd. (Industry)
Responsible Party: Dr. Adrian Frentzel, Mepha Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIT 001-2006
Record Dates: First submitted 2010-03-15; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Urinary Tract Infection
Keywords: urinary tract infection; nitrofurantoin
MeSH Terms: conditions — Urinary Tract Infections | interventions — Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitrofurantoin (Experimental): Adult patients with a microbiologically confirmed uncomplicated urinary tract infection
  Interventions: Drug: Nitrofurantoin

INTERVENTIONS:
Drug: Nitrofurantoin — 100 mg retard capsules to be taken twice daily for seven days
  Other Names: Uvamin retard

SUMMARY:
The study aims to investigate bacteriological efficacy of a nitrofurantoin formulation given twice daily for seven days in the treatment of adult patients with microbiologically confirmed uncomplicated urinary tract infection.

Additional study objectives are to evaluate clinical efficacy as well as safety and tolerability of the nitrofurantoin formulation.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women and men aged above 18 years old
* presence of ≥ 2 signs or symptoms suggestive of a UTI (dysuria, urinary frequency, urgency, suprapubic pain) with onset 10 days before enrollment
* asymptomatic patients with available positive urine culture
* pyuria defined as positive leucocyte esterase (LE) test with any color change after two minutes
* collection of clean-voided midstream urine sample for culture and susceptibility testing to confirm bacteriuria
* normal renal function (defined as blood creatinine < 1.4 mg/100 ml)
* able to take oral medication on an outpatient basis
* written informed consent before enrollment

Exclusion Criteria:

* suspicion of complicated UTI (presence of fever above 38°C, flank pain, known urologic structural abnormality) or prostatitis
* negative urine dipslide results (uropathogen < 100000 CFU (colony-forming units)/mL) or presence of nitrofurantoin resistant isolate uropathogens or mixed cultures of more than two isolates
* symptoms of UTI within the past 4 weeks
* evidence of predisposing factor to UTI (e.g. calculi, stricture, primary renal disease like polycystic renal diseases and neurogenic bladder)
* medical history of anaemia, complicated diabetes mellitus, peripheral neuropathy, vitamin B deficiency, renal insufficiency, other significant renal, hepatic or lung diseases
* medical history of glucose-6-phosphate dehydrogenase deficiency (G6PD)
* electrolytes disorders
* pregnant, breast-feeding women or not using medically accepted, effective method of birth control
* history of nitrofurantoin hypersensitivity
* use of systemic bacteriological agent within 48 hours before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of bacteriological efficacy | after 12-42 days
  Bacteriological efficacy is assessed by number and type of isolates in a clean-void midstream urine sample.

SECONDARY OUTCOMES:
Evaluation of clinical efficacy | after 12-42 days
  Clinical efficacy is assessed by the disappearance/improvement of clinical symptoms (dysuria, frequency, urgency, suprapubic pain).
Evaluation of safety and tolerability | 1-42 days
  Safety and tolerability of the nitrofurantoin formulation is assessed during whole duration of study by monitoring all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Mendoza Valdes, MD, Principal Investigator — Cif Biotec, Medical Sur
Locations (1):
- Cif Biotec, Medica Sur, Mexico City, Mexico